CLINICAL TRIAL: NCT07289789
Title: Comparative Effects of Buteyko Versus Pilates Breathing Combined With McKenzie Neck Exercises on Lung Function and Chest Expansion in Asthmatic Patients With Forward Head Posture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2025/94
Record Dates: First submitted 2025-09-12; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Asthma
Keywords: Breathing exercises; Respiratory Function Test; Chest Expansion; Mckenzie Neck Exercises
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- McKenzie neck exercises with Pilates-based breathing (Experimental): Participants in this group will perform McKenzie neck exercises in combination with Pilates-based breathing techniques, along with their usual pharmacological management for asthma. The program will run for 4 weeks with progressive intensity. McKenzie exercises will start with 5 repetitions per exercise in Weeks 1-2 and progress to 10 repetitions in Weeks 3-4. Pilates breathing will begin with 2 sets of 10 repetitions in Weeks 1-2, progress to 3 sets in Week 3, and 4 sets in Week 4.
  Interventions: Procedure: Pilates Breathing Combined with McKenzie Neck Exercises
- McKenzie neck exercises with Buteyko breathing technique (Experimental): Participants in this group will perform McKenzie neck exercises in combination with Buteyko breathing techniques, along with their usual pharmacological management for asthma. The program will run for 4 weeks with progressive intensity. McKenzie exercises will start with 5 repetitions per exercise in Weeks 1-2 and progress to 10 repetitions in Weeks 3-4. Buteyko breathing will begin with 2 sets of 10 repetitions in Weeks 1-2, progress to 3 sets in Week 3, and 4 sets in Week 4.
  Interventions: Procedure: McKenzie Neck Exercises with Buteyko Breathing

INTERVENTIONS:
Procedure: Pilates Breathing Combined with McKenzie Neck Exercises — Participants in this group will undergo a four-week intervention program combining McKenzie neck exercises with Pilates-based breathing techniques. The McKenzie exercises will be performed at an intensity of five repetitions per exercise during the first two weeks, progressing to ten repetitions per exercise in the third and fourth weeks. Pilates breathing will begin with two sets of ten repetitions in the first and second weeks, progress to three sets of ten repetitions in the third week, and further increase to four sets of ten repetitions in the fourth week. The intervention will be carried out three days per week on alternate days.
  Arms: McKenzie neck exercises with Pilates-based breathing
Procedure: McKenzie Neck Exercises with Buteyko Breathing — Participants in this group will undergo a four-week intervention program combining McKenzie neck exercises with Pilates-based breathing techniques. The McKenzie exercises will be performed at an intensity of five repetitions per exercise during the first two weeks, progressing to ten repetitions per exercise in the third and fourth weeks. Pilates breathing will begin with two sets of ten repetitions in the first and second weeks, progress to three sets of ten repetitions in the third week, and further increase to four sets of ten repetitions in the fourth week. The intervention will be carried out three days per week on alternate days
  Arms: McKenzie neck exercises with Buteyko breathing technique

SUMMARY:
Asthma is characterized by airway inflammation and hyperinflation that flattens the diaphragm and increases reliance on accessory neck muscles. Chronic overuse shortens these muscles and promotes forward head posture (FHP), which in turn compromises rib-cage motion and respiratory mechanics. Correcting FHP alongside breathing retraining may therefore improve lung function and symptoms in asthma. This interventional, parallel-group study investigates the combined effects of McKenzie neck exercises with two different breathing approaches on lung function, chest expansion, posture, and quality of life in adults with asthma. Participants are allocated to two groups for a 4-week program: Group A performs McKenzie neck exercises plus Pilates-based breathing; Group B performs McKenzie neck exercises plus Buteyko breathing.

DETAILED DESCRIPTION:
Asthma is a chronic inflammatory condition characterized by airway narrowing, hyperinflation, and increased airway resistance. Over time, these changes flatten the diaphragm, leading to reduced efficiency of the primary respiratory muscle. As a compensatory mechanism, asthmatic patients rely heavily on accessory muscles, particularly the sternocleidomastoid and scalene muscles. Prolonged overuse of these muscles contributes to shortening, tightness, and altered biomechanics of the cervical region, resulting in forward head posture (FHP). FHP negatively influences respiratory mechanics by reducing rib cage mobility, altering muscle recruitment patterns, and impairing effective exhalation. It is also associated with musculoskeletal discomfort and cervical spine stress, which further compound the challenges faced by asthmatic individuals.

Correcting FHP is therefore an important therapeutic target. Evidence suggests that restoring cervical alignment improves lung function parameters and breathing mechanics in patients with asthma. McKenzie neck exercises are a widely recognized approach for postural correction. These exercises aim to normalize cervical spine position, reduce stress on accessory muscles, and promote improved head and neck alignment. By addressing postural deviations, McKenzie exercises may indirectly enhance diaphragmatic function and overall ventilatory efficiency.

Breathing retraining techniques such as Pilates breathing and Buteyko breathing have also been shown to provide benefits for patients with asthma. Pilates-based breathing emphasizes controlled inhalation and exhalation with engagement of the diaphragm and rib cage expansion, promoting better respiratory coordination and relaxation. Buteyko breathing, in contrast, focuses on reducing hyperventilation and breath-holding techniques to optimize carbon dioxide levels and minimize airway irritation. Both methods target abnormal breathing patterns commonly found in asthma but through different mechanisms. This study is designed to examine the combined effect of postural correction and breathing retraining. Participants are randomly allocated into two groups, both receiving McKenzie neck exercises but paired with different breathing methods. Group A performs McKenzie exercises alongside Pilates-based breathing, while Group B combines McKenzie exercises with Buteyko breathing.

ELIGIBILITY:
Inclusion Criteria:

* Age group 18-40years
* Both males and females
* Individuals clinically diagnosed with asthma that is well controlled (Level 1 and Level 2) with FHP
* Not participated in any structured exercise regime for improving lung function during the past 6 months.
* Individuals well tolerated with a current exercise plan of combination exercises. (Buteyko breathing/Pilate breathing and McKenzie neck exercises

Exclusion Criteria:

* -Level 3 and 4 asthma or status asthmatics.
* Any congenital deformity of the chest wall
* Any active infections like fever, TB
* Those with any contraindication to exercise testing or training.
* Recent history of any chest wall trauma
* Any abdominal or cardio thoracic surgery
* Any psychiatric illness
* Unstable Cardiopulmonary disease i.e. unstable angina, heart failure, recent MI.
* Unstable hemodynamic parameters (arterial pressure >140mmhg systolic and >90mmhg for diastolic
* Pregnancy
* Previous or parallel participation in interventional programs.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Chest Expansion | 4 weeks
  Description: Chest expansion will be measured in centimeters using a standard measuring tape at the level of the 4th intercostal space.
Lung Functions | 04 weeks
  Lung function will be assessed using a spirometer. The parameters recorded will be FEV1 (Forced Expiratory Volume in 1 second), FVC (Forced Vital Capacity) and FEV1/FVC ratio.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, 44000, Islamabad, Pakistan